CLINICAL TRIAL: NCT06158373
Title: The Effect of Mother's Massage and Safe Swaddling on Bonding, Self-effıcacy and Vital Signs in Infants Undergoing Cardiovascular Surgery
Brief Title: Bonding, Self-effıcacy and Vital Signs in Infants Undergoing Cardiovascular Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Sirin Celik, Supervisor : Assoc. Prof. Dr., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SCelik; İlkay Güngör Satılmış (Registry Identifier: igungorsatilmis)
Record Dates: First submitted 2023-07-26; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Mother-Infant Interaction
Keywords: maternal; infant massage; safe swaddling; touching; congenital heart disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental design with pretest posttest control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Infant Massage Group (Experimental): infant massage
  Interventions: Other: infant massage practice
- Safe Swaddling Group (Experimental): safe swaddling
  Interventions: Other: Safe Swaddling
- Control Group (Sham Comparator): control group
  Interventions: Other: Control

INTERVENTIONS:
Other: infant massage practice — infant massage practice
  Arms: Infant Massage Group
Other: Safe Swaddling — Safe Swaddling
  Arms: Safe Swaddling Group
Other: Control — Control
  Arms: Control Group

SUMMARY:
Congenital heart diseases, the most common type of congenital anomalies, which affect approximately 3% of all live births and are the second most common cause of death in infants, are associated with 7% of all neonatal deaths. Among the interventions that can be applied with family-centered care of newborns followed in the intensive care unit, infant massage and safe wrapping are suggested interventions for mother-infant bonding and parental self-efficacy through the infant's sense of touch.

Objective: The aim of this study was to increase mother-infant attachment, increase the self-efficacy of the mother by taking an active role in baby care, reduce the baby's pain and stabilize vital signs, and increase the adaptation of the baby and the mother to the process and reduce the hospitalization day.

In this study, it was aimed to evaluate the effects of maternal massage and safe swaddling on attachment, self-efficacy, and vital signs of the infant in infants undergoing cardiovascular surgery (CVC).

The sample of the study, which was conducted in an experimental design with a pre-test-post-test control group, consisted of 36 infants and their mothers who had CVC between December 2020 and January 2022 and were hospitalized in the intensive care unit. Infant massage (n:12), safe swaddling (n:12) and control group (n:12) mothers were determined by computerized randomization. After the mother-infant pre-assessment questionnaire, Parental Self-Efficacy Scale (PSES) Scale, and Maternal Attachment Inventory (MAI) pre-tests were applied to the mothers, infant massage and safe swaddling instruction were given to the mothers. The hemodynamic findings of the infant were recorded before, during and after the practices. Post-tests were applied before hospital discharge.

DETAILED DESCRIPTION:
Of the 130 million children born in the world each year, four million die in the neonatal stage. Congenital heart disease (CHD) is a serious congenital anomaly that can be seen at a rate of 5-8 per 1000 live births and is associated with 7% of all neonatal deaths (Aykan et al., 2022; Ertürk, 2016). Although pediatric cardiology and pediatric cardiovascular surgery have advanced, current data show that 21% of infants with congenital heart disease still die in the first month and 40% die due to congenital malformations (Beider et al., 2010). Early diagnosis of CHD, which is difficult to diagnose due to hemodynamic difference, and planning the treatment are important in terms of reducing morbidity and mortality in children (Bulut et al., 2012). While most of the babies with severe heart disease die in the first weeks of their lives, 25% of them need surgical intervention in the first week of their life (Özkan et al., 2010).

Preterm and term newborns, who have to spend the first week of their lives in neonatal intensive care units, are exposed to many invasive procedures (2-3 or 8-10 times a day) and experience pain and stress for different reasons. The pain experienced by the baby can prevent his behavior, family-baby interaction, and the baby's adaptation to the outside world, as well as cause changes in the development of the brain and senses, and growth is negatively affected (Derebent, 2006). By maintaining the balance between medical interventions and good primary care, babies' stress, pain and anxiety symptoms should be reduced. Easy-to-apply, low-cost non-pharmacological methods can be effective alone in pain caused by small invasive interventions; It has been reported that when used together with pharmacological methods, they increase the effectiveness of drugs (Şaduman, 2011).

The mother, whose baby is in the intensive care unit, has difficulties in establishing a close relationship with her child, and the mother's anxiety makes the attachment process more difficult. Effective nursing interventions to meet the needs of parents; helping parents to understand the infant's reactions, expressing their fears and expectations, actively listening to them, answering questions honestly, informing the parent about the treatment plan and program. It is also a nurse's responsibility to ensure mother-child interaction by enabling the mother to participate more in the care of the child (Özyazıcıoğlu, 2009). Increasing maternal experiences is important in mother-infant interaction. The most important component of these interventions is that intensive care nurses help the mother to be a good observer in evaluating her behavior in order to increase the mother's self-confidence in taking care of the baby and to strengthen her better relationship with her baby. The goal is primarily to ensure that the mother perceives her baby positively. Then, it is to give the mother the opportunity to touch, hold, care and observe her baby and to support her to give sensitive and positive reactions to her reactions to environmental stimuli. Thus, the mother's self-confidence, her ability to read the baby's reactions and her ability to meet the baby's needs are increased (Aras et al., 2013). The most commonly used non-pharmacological techniques in the care of these babies are various techniques and therapies such as reducing environmental stimuli, individualized developmental care and evaluation program of the newborn, music therapy, breastfeeding, supporting non-nutritive sucking, giving sweet solution, skin-to-skin contact, changing position, hugging, kangaroo care, massage therapy and wrapping. These techniques and therapies have an improving effect on cardiovascular and skeletal muscle functions (Beider et al., 2010; Yıldız, 2017).

The sense of touch is very important in the child's perception of his environment, especially in the newborn and infancy period. The baby communicates and recognizes his environment through the sense of touch. Appropriate stimulation of the sense of touch supports psychosocial development. Baby massage is a simple, inexpensive and effective technique that is beneficial for baby development. Baby massage is a new practice in our country, which many families are interested in, both for this reason and because it allows parents to freely apply it to their babies. Touch is proof of love. The creation of mother-father-infant interaction and the development of healthy attachment affect the development of the baby and his whole life. The family's loving attachment to the baby is the most important factor that accelerates its healthy growth and development. Massage; It is the mechanical and nervous stimulation of the skin, subcutaneous adipose tissue, muscles, internal organs, metabolism, circulation and lymph system for therapeutic and/or protective purposes. Many positive effects such as providing relaxation, reducing painful muscle tensions, relieving sleep problems and pain, improving self-esteem in individuals with physical disorders and terminal illness, and managing mental health problems can be achieved with massage application (Gürol, 2010). In addition, baby massage is between mother and baby.

ELIGIBILITY:
Inclusion Criteria:

* Born term,
* Those who have undergone CVS surgery and sternatomy
* Pediatric CVD intensive care unit patients
* Extubated
* Watched accompanied by his mother
* Can be breastfed by his mother
* Can be fed enterally
* No arrhythmia
* Clotting factors are within normal limits
* Baby and mother with 'Not at Risk' or PCR result 'Negative'
* Babies whose mothers accept the training and practice within the scope of the research.

Exclusion Criteria

* Those with 'Risky' or PCR result 'Positive' baby and mother during follow-up
* Sudden weight loss or acute gastrointestinal system problems
* Babies who are at risk of bleeding and cannot feed (with chylothorax etc.)
* Extubated babies with risk of reintubation and respiratory distress
* Babies whose mothers leave them for various reasons.

Ages: 3 Months to 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Safe swaddling method and Pain Score | "until discharge from intensive care" or "4 to 86 day"
  The pain score of infants who have undergone cardiovascular surgery and whose mothers apply safe swaddling method is lower than the control group.
Infant massage method and Pain Score | "until discharge from intensive care" or "4 to 86 day"
  Infants who have undergone cardiovascular surgery who are given infant massage by their mothers have lower pain scores than the control group.
Safe swaddling method and body temperature | "until discharge from intensive care" or "between 36,6-37,5 degrees"
  Body temperature is infants who have undergone cardiovascular surgery and whose mothers applied safe swaddling are more stable compared to the control group.
Safe swaddling method and body temperature | "until discharge from intensive care" and "between 36,6-37,5 degrees"
  Body temperature is infants who have undergone cardiovascular surgery and whose mothers applied safe swaddling are more stable compared to the control group.
Safe swaddling method and respiratory rate | "until discharge from intensive care" and " between 30-60 times per minute"
  Respiratory rate is infants who have undergone cardiovascular surgery and whose mothers applied safe swaddling are more stable compared to the control group.
Infant massage method and respiratory rate | "until discharge from intensive care" and " between 30-60 times per minute"
  Respiratory rate is infants who have undergone cardiovascular surgery who are given infant massage by their mothers are more stable compared to the control group.
Safe swaddling method and mother-infant attachment | "until discharge from intensive care" or "4 to 86 day"
  The mother-infant attachment of mothers who apply safe swaddling method to their infants who have undergone cardiovascular surgery is higher than the control group.

SECONDARY OUTCOMES:
Infant massage method and mother-infant attachment | "until discharge from intensive care" or "4 to 86 day"
  Mothers who apply infant massage to their infants who have undergone cardiovascular surgery have higher mother-infant attachment than the control group.
Safe swaddling method and self-efficacy | "until discharge from intensive care" or "4 to 86 day"
  The self-efficacy of mothers who apply safe swaddling method to their infants who have undergone cardiovascular surgery is higher than the control group.
Infant massage method and self-efficacy | "until discharge from intensive care" or "4 to 86 day"
  The self-efficacy of mothers who apply infant massage to their infants who have undergone cardiovascular surgery is higher than the control group.

OTHER OUTCOMES:
Infant massage method and sleep duration | "until discharge from intensive care" or "30 minutes to 2 hour"
  Sleep duration is longer in infants who receive infant massage compared to the control group.
Safe swaddling and hospitalization day | "until discharge from intensive care" or "4 to 86 day"
  The duration of intensive care unit hospitalization is less in infants who are applied safe swaddling method compared to the control group.
Infant massage method and hospitalization day | "until discharge from intensive care" or "4 to 86 day"
  The duration of intensive care hospitalization is less in the infants who received infant massage compared to the control group.
Safe swaddling and Sleep duration | "until discharge from intensive care" or "30 minutes to 2 hour"
  Sleep duration is longer in the babies who received safe swaddling method compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: İlkay Gungor Satilmis, Doc.Dr., Study Director — İstanbul University-Cerrahpaşa
Locations (1):
- Sirin Celik, Maltepe, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Afand N, Keshavarz M, Fatemi NS, Montazeri A. Effects of infant massage on state anxiety in mothers of preterm infants prior to hospital discharge. J Clin Nurs. 2017 Jul;26(13-14):1887-1892. doi: 10.1111/jocn.13498. Epub 2017 Mar 24. PMID 27486850
- [Background] Beider S, Boulanger KT, Joshi M, Pan YP, Chang RK. Measuring the effects of massage on exercise performance and cardiopulmonary response in children with and without heart disease: a pilot study. Int J Ther Massage Bodywork. 2010 Sep 28;3(3):12-6. doi: 10.3822/ijtmb.v3i3.86. PMID 21589710
- [Background] Field T, Gonzalez G, Diego M, Mindell J. Mothers massaging their newborns with lotion versus no lotion enhances mothers' and newborns' sleep. Infant Behav Dev. 2016 Nov;45(Pt A):31-37. doi: 10.1016/j.infbeh.2016.08.004. Epub 2016 Sep 3. PMID 27599170
- [Background] Vicente S, Verissimo M, Diniz E. Infant massage improves attitudes toward childbearing, maternal satisfaction and pleasure in parenting. Infant Behav Dev. 2017 Nov;49:114-119. doi: 10.1016/j.infbeh.2017.08.006. Epub 2017 Sep 1. PMID 28866286
- [Background] Ferentzi H, Rippe RCA, Latour JM, Schubert S, Girch A, Jonebratt Stocker M, Pfitzer C, Photiadis J, Sandica E, Berger F, Schmitt KRL. Family-Centered Care at Pediatric Cardiac Intensive Care Units in Germany and the Relationship With Parent and Infant Well-Being: A Study Protocol. Front Pediatr. 2021 Aug 12;9:666904. doi: 10.3389/fped.2021.666904. eCollection 2021. PMID 34458208
- [Background] Re JM, Dean S, Mullaert J, Guedeney A, Menahem S. Maternal Distress and Infant Social Withdrawal (ADBB) Following Infant Cardiac Surgery for Congenital Heart Disease. World J Pediatr Congenit Heart Surg. 2018 Nov;9(6):624-637. doi: 10.1177/2150135118788788. PMID 30322360
- [Background] Kasparian NA, Kan JM, Sood E, Wray J, Pincus HA, Newburger JW. Mental health care for parents of babies with congenital heart disease during intensive care unit admission: Systematic review and statement of best practice. Early Hum Dev. 2019 Dec;139:104837. doi: 10.1016/j.earlhumdev.2019.104837. Epub 2019 Aug 24. PMID 31455569
- [Background] Gaskin K, Kennedy F. Care of infants, children and adults with congenital heart disease. Nurs Stand. 2019 Jul 26;34(8):37-42. doi: 10.7748/ns.2019.e11405. PMID 31468777
- [Background] Bowlby J. Attachment and loss: retrospect and prospect. Am J Orthopsychiatry. 1982 Oct;52(4):664-678. doi: 10.1111/j.1939-0025.1982.tb01456.x. No abstract available. PMID 7148988
- [Background] Wittkowski A, Garrett C, Calam R, Weisberg D. Self-Report Measures of Parental Self-Efficacy: A Systematic Review of the Current Literature. J Child Fam Stud. 2017;26(11):2960-2978. doi: 10.1007/s10826-017-0830-5. Epub 2017 Jul 6. PMID 29081640
- [Background] Pados BF, McGlothen-Bell K. Benefits of Infant Massage for Infants and Parents in the NICU. Nurs Womens Health. 2019 Jun;23(3):265-271. doi: 10.1016/j.nwh.2019.03.004. Epub 2019 May 3. PMID 31059673
- [Background] Serrano MS, Doren FM, Wilson L. Teaching Chilean mothers to massage their full-term infants: effects on maternal breast-feeding and infant weight gain at age 2 and 4 months. J Perinat Neonatal Nurs. 2010 Apr-Jun;24(2):172-81. doi: 10.1097/JPN.0b013e3181db5377. PMID 20442614
- [Background] Field T. Massage therapy research review. Complement Ther Clin Pract. 2014 Nov;20(4):224-9. doi: 10.1016/j.ctcp.2014.07.002. Epub 2014 Aug 1. PMID 25172313
- [Background] Pease AS, Fleming PJ, Hauck FR, Moon RY, Horne RS, L'Hoir MP, Ponsonby AL, Blair PS. Swaddling and the Risk of Sudden Infant Death Syndrome: A Meta-analysis. Pediatrics. 2016 Jun;137(6):e20153275. doi: 10.1542/peds.2015-3275. Epub 2016 May 9. PMID 27244847
- [Background] Barry ES. Co-sleeping as a proximal context for infant development: The importance of physical touch. Infant Behav Dev. 2019 Nov;57:101385. doi: 10.1016/j.infbeh.2019.101385. Epub 2019 Oct 23. PMID 31655427
- [Background] Dixley A, Ball HL. The effect of swaddling on infant sleep and arousal: A systematic review and narrative synthesis. Front Pediatr. 2022 Nov 30;10:1000180. doi: 10.3389/fped.2022.1000180. eCollection 2022. PMID 36533224
- [Background] Heo YJ, Oh WO. The effectiveness of a parent participation improvement program for parents on partnership, attachment infant growth in a neonatal intensive care unit: A randomized controlled trial. Int J Nurs Stud. 2019 Jul;95:19-27. doi: 10.1016/j.ijnurstu.2019.03.018. Epub 2019 Apr 2. PMID 31005676
- [Background] Golfenshtein N, Hanlon AL, Deatrick JA, Medoff-Cooper B. Parenting stress trajectories during infancy in infants with congenital heart disease: Comparison of single-ventricle and biventricular heart physiology. Congenit Heart Dis. 2019 Nov;14(6):1113-1122. doi: 10.1111/chd.12858. Epub 2019 Oct 27. PMID 31657114
- [Background] McClung N, Glidewell J, Farr SL. Financial burdens and mental health needs in families of children with congenital heart disease. Congenit Heart Dis. 2018 Jul;13(4):554-562. doi: 10.1111/chd.12605. Epub 2018 Apr 6. PMID 29624879
- [Background] Elgersma KM, McKechnie AC, Schorr EN, Shah KM, Trebilcock AL, Ramel SE, Ambrose MB, Swanson NM, Sommerness SA, Spatz DL. The Impact of Human Milk on Outcomes for Infants with Congenital Heart Disease: A Systematic Review. Breastfeed Med. 2022 May;17(5):393-411. doi: 10.1089/bfm.2021.0334. Epub 2022 Feb 15. PMID 35167760
- [Background] Jin X, Ni W, Wang G, Wu Q, Zhang J, Li G, Jiao N, Chen W, Liu Q, Gao L, Xing Q. Incidence and risk factors of congenital heart disease in Qingdao: a prospective cohort study. BMC Public Health. 2021 Jun 2;21(1):1044. doi: 10.1186/s12889-021-11034-x. PMID 34078335
- [Background] Mosiman W, Pile D. Emerging therapies in pediatric pain management. J Infus Nurs. 2013 Mar-Apr;36(2):98-106. doi: 10.1097/NAN.0b013e318282a8a5. PMID 23455971
- [Background] Fratellone PM, Steinfeld L, Coplan NL. Exercise and congenital heart disease. Am Heart J. 1994 Jun;127(6):1676-80. doi: 10.1016/0002-8703(94)90425-1. No abstract available. PMID 8198016
- [Background] Peterson JK. Supporting Optimal Neurodevelopmental Outcomes in Infants and Children With Congenital Heart Disease. Crit Care Nurse. 2018 Jun;38(3):68-74. doi: 10.4037/ccn2018514. PMID 29858197
- [Background] Kelly BA, Irigoyen MM, Pomerantz SC, Mondesir M, Isaza-Brando N. Swaddling and Infant Sleeping Practices. J Community Health. 2017 Feb;42(1):10-14. doi: 10.1007/s10900-016-0219-1. PMID 27393144
- [Background] van Sleuwen BE, Engelberts AC, Boere-Boonekamp MM, Kuis W, Schulpen TW, L'Hoir MP. Swaddling: a systematic review. Pediatrics. 2007 Oct;120(4):e1097-106. doi: 10.1542/peds.2006-2083. PMID 17908730
- [Background] Fang Y, Boelens M, Windhorst DA, Raat H, van Grieken A. Factors associated with parenting self-efficacy: A systematic review. J Adv Nurs. 2021 Jun;77(6):2641-2661. doi: 10.1111/jan.14767. Epub 2021 Feb 15. PMID 33590585
- [Background] Vance AJ, Pan W, Malcolm WH, Brandon DH. Development of parenting self-efficacy in mothers of high-risk infants. Early Hum Dev. 2020 Feb;141:104946. doi: 10.1016/j.earlhumdev.2019.104946. Epub 2019 Dec 31. PMID 31901656
- [Background] Harrison TM, Brown R, Duffey T, Frey C, Bailey J, Nist MD, Renner L, Fitch J. Effects of Massage on Postoperative Pain in Infants With Complex Congenital Heart Disease. Nurs Res. 2020 Sep/Oct;69(5S Suppl 1):S36-S46. doi: 10.1097/NNR.0000000000000459. PMID 32858717
- [Background] Jordan B, Franich-Ray C, Albert N, Anderson V, Northam E, Cochrane A, Menahem S. Early mother-infant relationships after cardiac surgery in infancy. Arch Dis Child. 2014 Jul;99(7):641-5. doi: 10.1136/archdischild-2012-303488. Epub 2014 Mar 17. PMID 24636955
- [Background] Shoghi M, Sohrabi S, Rasouli M. The Effects of Massage by Mothers on Mother-Infant Attachment. Altern Ther Health Med. 2018 May;24(3):34-39. PMID 29101776
- [Background] Kohlhoff J, Barnett B. Parenting self-efficacy: links with maternal depression, infant behaviour and adult attachment. Early Hum Dev. 2013 Apr;89(4):249-56. doi: 10.1016/j.earlhumdev.2013.01.008. Epub 2013 Feb 8. PMID 23398731
- [Background] Bernard NK, Bogat GA, Kashy DA, Lonstein JS, Levendosky AA. Prenatal and postnatal intimate partner violence, depression, and infant-mother touch. Infant Behav Dev. 2022 May;67:101703. doi: 10.1016/j.infbeh.2022.101703. Epub 2022 Feb 25. PMID 35220177
- [Background] Crucianelli L, Wheatley L, Filippetti ML, Jenkinson PM, Kirk E, Fotopoulou AK. The mindedness of maternal touch: An investigation of maternal mind-mindedness and mother-infant touch interactions. Dev Cogn Neurosci. 2019 Feb;35:47-56. doi: 10.1016/j.dcn.2018.01.010. Epub 2018 Jan 31. PMID 29402735
- [Background] Nelson AM. Risks and Benefits of Swaddling Healthy Infants: An Integrative Review. MCN Am J Matern Child Nurs. 2017 Jul/Aug;42(4):216-225. doi: 10.1097/NMC.0000000000000344. PMID 28394766
- [Background] Rudnicki J, Boberski M, Butrymowicz E, Niedbalski P, Ogniewski P, Niedbalski M, Niedbalski Z, Podraza W, Podraza H. Recording of amplitude-integrated electroencephalography, oxygen saturation, pulse rate, and cerebral blood flow during massage of premature infants. Am J Perinatol. 2012 Aug;29(7):561-6. doi: 10.1055/s-0032-1310529. Epub 2012 Apr 11. PMID 22495901
- [Background] Rana D, Garde K, Elabiad MT, Pourcyrous M. Whole body massage for newborns: A report on non-invasive methodology for neonatal opioid withdrawal syndrome. J Neonatal Perinatal Med. 2022;15(3):559-565. doi: 10.3233/NPM-220989. PMID 35599503
- [Background] Nyaga E, Esamai F, Kyololo O. Effect of massage therapy on preterm neonate's body temperature. Afr Health Sci. 2021 Sep;21(3):1334-1339. doi: 10.4314/ahs.v21i3.44. PMID 35222598
- [Background] Chanvorachote P, Jirachotdecho K, Suksumek N. A Randomized Controlled Trial of Evaluating the Efficacy of Alternative Swaddles for Body Temperature Control of Newborns. In Vivo. 2022 Jul-Aug;36(4):1966-1970. doi: 10.21873/invivo.12919. PMID 35738617